CLINICAL TRIAL: NCT02013739
Title: Description of Insulin Resistance and Explanatory Variables in Patients With Chronic Heart Failure
Brief Title: Description of Insulin Resistance in Patients With Chronic Heart Failure
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Bert Op't Eijnde, prof. dr., Hasselt University
Other Study IDs: 11.78/cardio11.13
Record Dates: First submitted 2013-12-08; First posted 2013-12-17 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with chronic heart failure: other
- Healthy volontiers: other

SUMMARY:
The purpose of this study is to describe insulin resistance in a general chronic heart failure population, in combination with muscle strength, body composition and cardiac function.

It is assumed that insulin resistance is increased in CHF patient, and that this is related to decreased muscle strength and decreased lean tissue mass.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic heart failure for at least 6 months,
* clinically stable (not hospitalized) for more than 3 months prior to the onset of the study,

Exclusion Criteria:

* glucose lowering medical therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with chronic heart failure
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance | day1
  glucose and insulin concentration measurements in blood during oral glucose tolerance test

SECONDARY OUTCOMES:
HbA1c, blood lipids, BNP | day 1
Muscle strength: maximal strength tested on a isokinetic dynamometer | Day 1
Body composition: dual energy x-ray absorptiometry | Day 1
cardiac function: echocardiography, retrospective from hospital files | retrospective
Health-related quality of life: MLHFQ and Eq5d | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Bert Op 't Eijnde, prof. dr., Principal Investigator — Hasselt University
Locations (1):
- Hasselt University, Hasselt, Limburg, Belgium